CLINICAL TRIAL: NCT01458080
Title: WEUSKOP5410: A Retrospective Observational Non-Interventional Nested Case Control Study to Evaluate the Risk for Thromboembolic Events Associated With Surgery and Eltrombopag Exposure in the ENABLE Studies
Brief Title: WEUSKOP5410: Observational Study in ENABLE Clinical Trials
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115885; EPI40664 (Other: GSK); WEUSKOP5410 (Other: GSK)
Record Dates: First submitted 2011-07-07; First posted 2011-10-24 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis C
Keywords: ENABLE; invasive procedures; Thrombocytopenia; Thromboembolic events; Eltrombopag; Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C; Thrombocytopenia; Thromboembolism | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients w/secondary thrombocytopenia related to hepatitis C: Patients w/secondary thrombocytopenia related to hepatitis C
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — eltrombopag

SUMMARY:
Hepatitis C Virus (HCV) is a leading cause of chronic liver disease (CLD) worldwide. Current mainstay of treatment is combination therapy with pegylated interferon and ribavarin. Thrombocytopenia as a treatment related adverse event or a complication of chronic liver disease often necessitates dose reduction and discontinuation in these patients. Revolade®/Promacta® (eltrombopag) is an oral second generation thrombopoietic growth factor in development for the treatment thrombocytopenia associated with various conditions, including secondary thrombocytopenia related to CLD and hepatitis C. In 2009 a phase III trial for CLD patients undergoing an elective invasive procedure (ELEVATE) was terminated early due to an imbalance of thromboembolic events (TEE) between the placebo and the eltrombopag arm. Currently, two global interventional Phase III trials (ENABLE 1 and ENABLE 2) are being conducted in approximately 1500 patients to evaluate the efficacy of eltrombopag in enabling HCV patients to achieve sustained viral response. Due to the similarities between the patient groups in ELEVATE and ENABLE, there is a concern that invasive procedures may influence the risk of TEE in the ENABLE population. This observational, non-interventional, retrospective, multicentre, nested case-control study will collect data from chart abstraction and medical record review to augment data from the ENABLE case report forms particularly with regards to invasive procedures. The study population includes cases and controls drawn from the ~1500 participants of the ENABLE trials. All eligible cases of TEE will be included in the study as cases. All other patients who participated in the ENABLE trials and did not experience a TEE, will be eligible to be selected as controls. Case report forms will be developed to enable standardized data capture. The Sponsor has contracted with the Clinical Research Organization, Outcome Sciences Inc to manage the study. ENABLE investigators will work with Outcome staff to obtain relevant information from the treating physician (e.g. surgeon) and the facility where the invasive procedure was performed (pre-operative tests, peri-operative course, diagnostic testing for TEE). Single point abstraction will be performed to obtain data from the medical record and from any additional data resources obtained by the investigator (e.g., operative note, anesthesia record). Analyses will be conducted using logistic regression models to estimate the risks. The primary objective of the study is to evaluate if there is an increased risk for TEE among patients who had an invasive procedure while exposed to eltrombopag (during the ENABLE trials).

ELIGIBILITY:
- The inclusion criteria for this case-control study was that the patients had to be participating in both the open-label phase and the randomization phase of any of ENABLE 1 or ENABLE 2 clinical trials.

Inclusion criteria for the ENABLE clinical trials included

* age>18 years
* evidence of chronic HCV infection
* candidates for peg-interferon and ribavirin combination antiviral therapy
* baseline platelet count of <75,000/µl
* no significant anemia or neutropenia.

Exclusion criteria for the ENABLE clinical trial included:

* non-responders to previous treatment with peg-interferon and ribavirin unless due to thrombocytopenia
* decompensated liver disease, e.g. Child-Pugh score >6 or history of ascites or hepatic encephalopathy or current evidence of ascites
* serious cardiac, cerebrovascular, or pulmonary disease
* documented history of clinically significant bleeding from oesophageal or gastric varices, haemoglobinopathies, e.g. sickle cell anemia, thalassemia major, history of arterial or venous thrombosis, hepatocellular carcinoma, Human Immunodeficiency Virus (HIV) or Hepatitis B infection
* any disease condition associated with active bleeding or requiring anticoagulation
* history of malignancy, history of alcohol/drug abuse or dependence within 6 months of the study start
* history of platelet clumping that prevents reliable measurement of platelet counts
* history of major organ transplantation with an existing functional graft
* evidence of portal vein thrombosis on abdominal imaging within 3 months of the baseline visit.

No additional exclusion criteria were applied to the case-control study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this study comprised all patients who participated in both the open-label phase and the randomization phase of any of ENABLE 1 or ENABLE 2 clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
diagnosis of a thromboembolic event during the study period. | The patients will be followed from the time of entry into the ENABLE 1 or ENABLE 2 clinical trial up until the index date, defined as the time of event for the case.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline